CLINICAL TRIAL: NCT06045650
Title: Relationship Between Oxytocin Level, Trust, and Attachment in Individuals With Borderline Personality Disorder
Status: Not yet recruiting | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Luba Leontieva, M.D./PhD, Director of Inpatient Unit, Associate Professor, Department of Psychiatry and Behavioral Sciences, State University of New York - Upstate Medical University
Other Study IDs: 2060971
Record Dates: First submitted 2023-09-07; First posted 2023-09-21 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Borderline Personality Disorder
Keywords: oxytocin; borderline personality disorder; trust-related behavior; attachment styles; childhood trauma; emotional sensitivity
MeSH Terms: conditions — Borderline Personality Disorder; Hypersensitivity | interventions — Childhood Trauma Questionnaire

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Participants with borderline personality disorder who meet the inclusion criteria
  Interventions: Other: baseline serum oxytocin levels; Other: Emotional Sensitivity test; Other: Neuro-economical game; Other: Childhood Trauma Questionnaire; Other: Relationships Questionnaire; Other: demographic questionnaire
- Controls: Participants without borderline personality disorder, who meet the inclusion criteria
  Interventions: Other: baseline serum oxytocin levels; Other: Emotional Sensitivity test; Other: Neuro-economical game; Other: Childhood Trauma Questionnaire; Other: Relationships Questionnaire; Other: demographic questionnaire

INTERVENTIONS:
Other: baseline serum oxytocin levels — Both cases and controls will be assessed for their baseline serum oxytocin levels
Other: Emotional Sensitivity test — To assess the level of emotional sensitivity in the participant
Other: Neuro-economical game — A game played to assess the trust-index of participants
Other: Childhood Trauma Questionnaire — to assess childhood trauma score
Other: Relationships Questionnaire — to assess attachment type
Other: demographic questionnaire — To obtain basic data on demographics

SUMMARY:
We aim to assess the baseline oxytocin levels in individuals with borderline personality disorder and correlate those levels with social behavior, and compare the results with controls.

Primary Hypothesis (H1):

There is a significant difference in trust-related behavior as measured by oxytocin (OXT) levels between borderline personality disorder (BPD) patients and healthy controls.

Secondary Hypotheses:

H2: The trust-related behavior in BPD patients is significantly influenced by their level of emotional sensitivity. Specifically, higher emotional sensitivity in BPD patients is associated with lower trust-related behavior and vice-versa.

H3: There is a significant correlation between trust-related behavior and childhood trauma in BPD patients. BPD patients with higher levels of reported childhood trauma will exhibit lower trust-related behavior compared to those with lower levels of trauma.

H4: Trust-related behavior in BPD patients varies depending on their attachment styles. Specifically, BPD patients with insecure attachment styles will exhibit lower trust-related behavior compared to those with secure attachment styles.

H5: There is a significant correlation between trust-related behavior and BPD severity. Patients with more severe BPD symptoms will exhibit lower trust-related behavior compared to those with less severe symptoms.

H6: The levels of OXT in BPD patients will significantly correlate with their reported levels of emotional sensitivity, childhood trauma, attachment styles, and BPD severity.

These hypotheses aim to address the complexities surrounding the modulation of trust-related behavior by oxytocin in BPD patients, taking into account various factors like emotional sensitivity, childhood adversity, attachment styles, and BPD severity. By testing these hypotheses, the study aims to provide a comprehensive understanding of the interplay between these factors in influencing trust-related behavior in BPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with borderline personality disorder will qualify as cases
* controls will be age, gender matched individuals without any psychiatric/mental health concerns

Exclusion Criteria:

* for all: pregnancy, hormonal or neurological disorders, and any kind of regular medication
* additional exclusion criteria for cases: a lifetime diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or significant neurological disease, current alcohol/ drug dependence
* for controls: MacLEan screening instrument for BPD will be used at the time of screening to exclude BPD diagnosis in controls

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: cases: individuals who are admitted to the inpatient psychiatry unit at a university hospital controls: healthy volunteers who volunteer to participate from the same city as the university hospital
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of Oxytocin levels and trust index | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided